CLINICAL TRIAL: NCT03595254
Title: Thrive-Montana: A Computerized Cognitive Behavior Therapy (cCBT) Program to Reduce Depression, Anxiety, Suicidal Ideation and Behaviors for Rural Montanans
Brief Title: Digital Cognitive Behavior Therapy Program for Suicide Prevention
Acronym: TM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Montana Department of Public Health and Human Services (Unknown)
Responsible Party: Principal Investigator, Mark B. Schure, Ph.D., Assistant Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSchure
Record Dates: First submitted 2018-06-29; First posted 2018-07-23 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Suicidal Ideation; Depression; Anxiety
MeSH Terms: conditions — Suicidal Ideation; Depression; Anxiety Disorders | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: randomized waitlist controlled trial (first ?? participants) Open trial (following ?? participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrive Intervention (Experimental): Online cognitive behavior therapy program
  Interventions: Behavioral: Thrive
- Waitlist Control (No Intervention): Wait 8 weeks before receiving program access

INTERVENTIONS:
Behavioral: Thrive — Computerized Cognitive Behavior Therapy program
  Other Names: Thrive-Montana
  Arms: Thrive Intervention

SUMMARY:
This study evaluates the efficacy of Thrive, a computerized cognitive behavior therapy program, to reduce depression and anxiety symptoms and to reduce suicidal thinking among adults. The first 450 participants will participate in a randomized waitlist controlled trial. The remaining 550 participants will be provided the program immediately upon enrolling

DETAILED DESCRIPTION:
The efficacy of Thrive has been studied among patient and community populations and has shown to effectively reduce depression and anxiety symptoms among adults with moderate to severe depression symptoms at baseline.

This study will examine whether Thrive can also reduce suicidal thinking for persons exhibiting at least moderate depression symptoms. The first phase of the study will implement a randomized waitlist controlled trial. The second phase of the study will examine the effects in a open trial. Outcome assessments will occur at baseline, 4- and 8-weeks (12- and 16-weeks for the waitlist group) with a 6-month follow-up assessment for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Montana resident
* 18+ years old
* Have regular access to broadband internet
* PHQ-9 score greater than 4

Exclusion Criteria:

* No Montana residency
* < 18 years old
* No broadband internet access
* PHQ-9 score less than 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Concise Health Risk Tracking | 2 Weeks
  Suicidal Thinking; Score range 7 (better) - 35(worse)

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Scale-7 | 2 Weeks
  Anxiety symptoms; Score range 0 (better) to 21 (worse)
Work and Social Adjustment Scale | 1 Year
  Functioning; Score range 0(better) - 40(worse)
Connor-Davidson Resilience Scale - Abbreviated Version | 1 month
  Resilience; score range 0 (worse) - 40(better)
Patient Health Questionnaire-9 | 2 Weeks
  Depression; Score range 0(better) - 27(worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No